CLINICAL TRIAL: NCT06873308
Title: Assessment of Infection Activity in Travelers and Migrants Diagnosed With Chronic Schistosomiasis: a Multicentric Prospective Cohort Study
Brief Title: Assessment of Infection Activity in Travelers and Migrants Diagnosed With Chronic Schistosomiasis
Acronym: SchistAct
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Collaborators: Leiden University Medical Center (LUMC) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-05
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Schistosomiasis
Keywords: schistosomiasis; chronic; diagnosis
MeSH Terms: conditions — Schistosomiasis; Bronchiolitis Obliterans Syndrome; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants (Other): All eligible participants identified as having chronic schistosomiasis according to site-specific diagnostic practice will have a standardized baseline clinical and laboratory assessment at enrollment that will include blood sampling for hematology, Schistosoma serology available at each site, and PCR for Schistosoma where available; urine sampling for microscopy, determination of hematuria as indirect markers of schistosomiasis morbidity, and Schistosoma PCR (where available) and POC-CCA urine strip assay (where available); and stool sampling for microscopy and PCR where available, and fecal occult blood as indirect markers of schistosomiasis morbidity. Serum (at least 1 mL leftover from routine diagnostics) will be sent to LUMC, Netherlands, where CAA will be determined with the UCP-LF CAA assay (dry format) designed for routine use.
  Interventions: Device: UCP-LF CAA assay

INTERVENTIONS:
Device: UCP-LF CAA assay — dry LF-CAA, or CAA

SUMMARY:
The primary objective of this clinical investigation is to determine the percentage of travelers and migrants diagnosed with chronic schistosomiasis according to site-specific diagnostic practice who have active infection at the time of evaluation (as assessed and classified by composite reference standards that integrate clinical, laboratory, and diagnostic features, such as microscopy, PCR (where available), POC-CCA (where available), and serum CAA results).

All subjects with chronic schistosomiasis according to site-specific diagnostic practice will have a standardized baseline clinical and laboratory evaluation at the time of evaluation that will include blood sampling for hematology, schistosome serology available at each site, and schistosome PCR where available; urine sampling for microscopy, determination of hematuria as an indirect marker of morbidity for schistosomiasis, and Schistosome PCR (where available), and urine strip testing POC-CCA (where available); and stool sampling for microscopy and PCR, where available, and fecal occult blood as indirect markers of schistosomiasis morbidity.

Composite reference standards will be used to assess and classify the activity of the infection. Organ-specific ultrasound and other tests will be left to the physician's decision, but results will also be collected.

Serum (at least 1 ml remaining from routine diagnostics) will be sent to LUMC, the Netherlands, where CAA will be determined with the UCP-LF CAA test designed for routine use.

Participants will be asked to sign an additional consent form, which is optional and not precluding enrollment in the study, to allow the remaining serum to be stored at LUMC for 15 years, to allow secondary research.

ELIGIBILITY:
Inclusion criteria

1. diagnosis of chronic schistosomiasis (>3 months after last potential exposure) according to site-specific diagnostic practice
2. signed informed consent (and assent for minors).

Exclusion criteria

1. age below 5 years;
2. exposure to praziquantel after the last potential exposure to schistosomes
3. acute infection, i.e. likely infection <3 months before presentation

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Active infection | Baseline
  Proportion of enrolled participants fulfilling the composite reference standards for active infection:
  * Microscopy (Positive/Negative)
  * PCR (Positive/Negative, if performed)
  * CAA (Positive/Negative)
  * Serology (Positive/Negative)

SECONDARY OUTCOMES:
CAA result | Baseline
  Number of enrolled participants with positive CAA result at inclusion compared to number of those fulfilling the composite reference standards active infection and of those positive by each separate diagnostic method
  * Microscopy (P/N)
  * PCR (P/N)
  * CAA (P/N)
  * Serology (P/N)
  * POC-CCA (P/N)
  * Signs/symptoms (eosinophilia (Y/N; eos/μL), hematuria (Y/N), fecal occult blood (Y/N), bladder mucosal lesions (Y/N, if ultrasound performed)

OTHER OUTCOMES:
CAA cure | At week 6 post-treatment
  Number of participants who will be CAA negative at week 6 post-treatment compared to number of participants fulfilling the definitions of cure and to number of negative results by each other separate diagnostic method.
  * Microscopy - viable eggs (P/N)
  * CAA (P/N)
  * Signs/symptoms (eosinophilia (Y/N; eos/μL), hematuria (Y/N), fecal occult blood (Y/N)

CONTACTS AND LOCATIONS:
Overall Officials: Federico Giovanni Gobbi, Principal Investigator — IRCCS Sacro Cuore Don Calabria
Locations (8):
- Institute of Tropical Medicine (ITM), Antwerp, Belgium
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany
- Italy (3):
  - IRCCS Policlinico Sant'Orsola, Bologna, BO
  - IRCCS Sacro Cuore Don Calabria, Negrar, VR
  - AOU Careggi, Florence
- Medical Microbiology & Infectious Diseases, Erasmus MC, Rotterdam, Netherlands
- Spain (2):
  - Tropical Medicine Unit of Hospital de Poniente, Almería
  - Vall d'Hebron University Hospital, Barcelona